CLINICAL TRIAL: NCT05158270
Title: Erector Spinae Plane Block for Postoperative Analgesia in Laparoscopic Cholecystectomy, is It a Promising Alternative Modality?
Brief Title: Erector Spinae Plane Block Versus Subcostal Anterior Quadratus Lumborum Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ashraf Torki, Lecturer of Anesthesia, Zagazig University, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB #9090
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Laparoscopic Cholecystectomy; Quadratus Lumborum Block; Erector Spinae Plane Block
Keywords: Laparoscopic cholecystectomy; Quadratus lumborum block; Erector spinae plane block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Computer-generated randomization numbers will be used to randomly assign patients into 3 groups using sealed opaque envelopes that will be randomly selected by each patient and contained a group number in which the patient was enrolled. Once enrolled in the study, patients will be randomly assigned into 3 groups;
  Group I (ESP Group): will receive US-guided ESPB. Group II (AQL Group): will receive US-guided AQLB. Group III (Control Group): will receive IV multimodal analgesia only.
  Both patients and data collector responsible for assessing outcomes will be blinded to group assignment (double-blinded clinical trial).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ultrasound Guided Erector Spinae Plane Block (Active Comparator): Patient will be placed in lateral decubitus position. By palpation of spinous processes starting from C7 downward, T7 spinous process will be located. Under complete aseptic precautions, linear probe of US machine will be placed in a transverse orientation at this level to identify tip of T7 transverse process (TP). By probe rotation into a longitudinal orientation, a parasagittal view will visualize skin and subcutaneous tissue, trapezius, and erector spinae (ES) muscle layers superficial to TPs. After local anesthetic (LA) infiltration, a 20 gauge spinal needle will be inserted in-plane and directed cranio-caudally until it contacts T7 TP. Target site for injection will be fascial plane deep to ES muscle. 1 mL saline will be injected to confirm correct needle-tip position by visualization of lifting of ES muscle off TP without distending the muscle and spreading cranio-caudally. 30 mL of 0.25% bupivacaine will be injected. Procedure will be performed bilaterally.
  Interventions: Procedure: Ultrasound Guided Erector spinae plane block
- Ultrasound Guided Subcostal Anterior Quadratus Lumborum Block (Active Comparator): Patients will be positioned lateral decubitus. A curvilinear 2-5 MHz ultrasound transducer (SonoSite S-Nerve, Bothell, WA) will be positioned posteriorly below the 12th rib in a parasagittal oblique plane at L1-2 level. The QL muscle was visualized and its point of insertion on the 12th rib identified. An 18-gauge Tuohy needle was advanced in the caudal-to-cranial direction between QL muscle and the psoas major muscle until a click could often be felt as the needle tip penetrated the anterior investing fascia of the QL muscle. After a negative aspiration, 30 mL of 0.25% bupivacaine was injected through the needle to help confirm the final needle tip position, anterior to the QL muscle at close proximity to the 12th rib.
  Interventions: Procedure: Ultrasound Guided Subcostal Anterior Quadratus Lumborum Block
- Intravenous Multimodal Analgesia (Other): Postoperative pain in the post-anesthesia care unit (PACU) and on the ward will be treated with a combination of IV multimodal analgesia in the form of Acetaminophen (15 mg/kg 4/day) and Ketorolac (0.5 mg/kg 3/day) using a fixed scheme. In addition, Nalpuphine, as 3 mg IV bolus at each dose, will be given when Numerical Rating Scale (NRS) ≥ 3. VAS will be assessed 5 - 10 min. after each opioid dose to assess the need for additional opioid doses.
  Interventions: Other: Intravenous Multimodal Analgesia

INTERVENTIONS:
Procedure: Ultrasound Guided Erector spinae plane block — Patient will be placed in lateral decubitus position. By palpation of spinous processes starting from C7 downward, T7 spinous process will be located. Under complete aseptic precautions, linear probe of US machine will be placed in a transverse orientation at this level to identify tip of T7 transverse process (TP). By probe rotation into a longitudinal orientation, a parasagittal view will visualize skin and subcutaneous tissue, trapezius, and erector spinae (ES) muscle layers superficial to TPs. After local anesthetic (LA) infiltration, a 20 gauge spinal needle will be inserted in-plane and directed cranio-caudally until it contacts T7 TP. Target site for injection will be fascial plane deep to ES muscle. 1 mL saline will be injected to confirm correct needle-tip position by visualization of lifting of ES muscle off TP without distending the muscle and spreading cranio-caudally. 20 - 30 mL of 0.25% bupivacaine will be injected. Procedure will be performed bilaterally.
  Arms: Ultrasound Guided Erector Spinae Plane Block
Procedure: Ultrasound Guided Subcostal Anterior Quadratus Lumborum Block — Patients will be positioned lateral decubitus. A curvilinear 2-5 MHz ultrasound transducer (SonoSite S-Nerve, Bothell, WA) will be positioned posteriorly below the 12th rib in a parasagittal oblique plane at L1-2 level. The QL muscle was visualized and its point of insertion on the 12th rib identified. An 18-gauge Tuohy needle was advanced in the caudal-to-cranial direction between QL muscle and the psoas major muscle until a click could often be felt as the needle tip penetrated the anterior investing fascia of the QL muscle. After a negative aspiration, 30 mL of 0.25% bupivacaine was injected through the needle to help confirm the final needle tip position, anterior to the QL muscle at close proximity to the 12th rib.
  Other Names: Ultrasound Guided Quadratus Lumborum Block
  Arms: Ultrasound Guided Subcostal Anterior Quadratus Lumborum Block
Other: Intravenous Multimodal Analgesia — Postoperative pain in the post-anesthesia care unit (PACU) and on the ward will be treated with a combination of IV multimodal analgesia in the form of Acetaminophen (15 mg/kg 4/day) and Ketorolac (0.5 mg/kg 3/day) using a fixed scheme. In addition, Nalpuphine, as 3 mg IV bolus at each dose, will be given when Numerical Rating Scale (NRS) ≥ 3. VAS will be assessed 5 - 10 min. after each opioid dose to assess the need for additional opioid doses.
  Arms: Intravenous Multimodal Analgesia

SUMMARY:
Adequate analgesic regimen is one of the most important key elements of Enhanced recovery after surgery (ERAS) protocols. The cornerstone of analgesia is multimodal analgesia combining local anesthetic (LA) techniques and trying to avoid parenteral opioids and their side effects. Subcostal approach to Anterior quadratus lumborum block (SAQLB), compared to other variants of quadratus lumborum blocks (QLBs), was associated with wider and longer sensory blockade, and provided somatic as well as visceral analgesia of the abdomen. The newly emerging, relatively easy erector spinae plane block (ESPB) provided excellent analgesia across a variety of surgical procedures and reduced opioid consumption. This motivated us to do this study to assess and compare the analgesic efficacy of ESPB versus SAQLB following laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Site of the Study: Zagazig university surgical hospitals.

Type of the Study: Prospective randomized double-blinded clinical trial.

Sample Size:

The sample size is calculated to be 27 for each group, assuming that the mean ± standard deviation of 24 hrs postoperative total opioid consumption among group of patients undergoing ESBP technique versus control group is 130 ± 88 and 201 ± 78, respectively. Assuming that US-guided SAQLB will be similar to ESBP technique in 24 hrs postoperative total opioid consumption. with confidence level of 95% and power of test 80%, with 10% drop out.

Withdrawal Criteria:

The patient has the right to withdraw from the study at any time without any negative consequences on medical or surgical treatment plan.

Randomization:

Computer-generated randomization numbers will be used to randomly assign patients into 3 groups using sealed opaque envelopes that will be randomly selected by each patient and contained a group number in which the patient was enrolled. Once enrolled in the study, patients will be randomly assigned into 3 groups;

Group I (ESP Group): will receive US-guided erector spinae plane block (ESPB). Group II (AQL Group): will receive US-guided subcostal anterior quadratus lumborum block (SAQLB).

Group III (Control Group): will receive intravenous (IV) multimodal analgesia only.

Clinician performing the blocks and patients will not be blinded, but investigators evaluating the outcomes will be blinded to the randomization to keep the data analysis unbiased.

Type of the Study: Prospective randomized double-blinded clinical trial.

Steps of Performance:

A. Intraoperative Management:

Preoperative Assessment:

All patients will be assessed by careful history taking, clinical examination and laboratory investigations. Laboratory work needed included; Complete blood count (CBC), biochemistry and coagulation profile. Other investigations (e.g., electrocardiography [ECG], echocardiography, and chest x-ray) will be done according to the patient's medical condition.

Preoperative Preparation:

The day before surgery, the purpose of this study, benefits from the block and possible complications that may occur will be explained clearly to the patient. After that, informed written consent will be obtained from him. Standard fasting guidelines will be also explained to the patients, i.e., no solid foods for 6 - 8 hrs (depending on fat content of the food) and no clear liquids for 2 hrs. Also, for aspiration prophylaxis, all patients will be instructed to take Erythromycin tablet 250 mg with Ranitidine tablet 150 mg, with 10 ml of water 2 hrs before procedure.

Premedication:

On arrival to the operating room, and after ensuring of working 18 gauge IV line, midazolam (2 mg) will be given IV for anxiolysis, then IV fluid drip will be started.

B. Intraoperative Management:

Intraoperative Monitoring:

Monitoring will be applied and maintained throughout the procedure, including 5- lead electrocardiogram (ECG), non-invasive arterial blood pressure, pulse oximeter, and capnography.

Hemodynamic parameters including heart rate (HR) and mean arterial blood pressure (MAP), will be recorded after receiving sedation (baseline data) and intraoperative immediately after induction, then every 5 minutes for 15 minutes, then every 15 minutes afterwards till the end of surgery.

General Anesthesia:

1. Induction and Intubation:

   Pre-oxygenation; will be done by asking the patient to take 8 vital capacity breaths of 100% O2 over one min. via a tightly fitting face-mask. Intravenous induction will be done using Fentanyl (1 µg/kg), Propofol (2 mg/kg) and Cis-atracurium (0.15 mg/kg). Mask ventilation will be done with 100% O2 for 3 min. until complete muscle paralysis. Endotracheal tube of suitable size will be used for tracheal intubation.
2. Immediately after Induction: Dexamethasone 8 mg IV will be given to all patients for prevention of postoperative nausea and vomiting (PONV).
3. Maintenance:

Anesthesia will be maintained with oxygen and 1.5% isoflurane. Additional doses of cis-atracurium (0.04 mg/kg) will be given when needed, guided by nerve stimulator. Volume-controlled mechanical ventilation will be used to maintain end-tidal carbon dioxide of 35-40 mmHg. Ventilator settings will be tidal volume 8 ml/kg and respiratory rate 10-15/min.

IV Fentanyl (0.5 - 1 mic/kg) will be given if MAP or HR increased 20% above baseline.

30 min. before the end of surgery, all patients will receive a combination of IV multimodal analgesia for postoperative pain control in the form of Acetaminophen (15 mg/kg), Ketorolac (0.5 mg/kg) and Nalbuphine (0.1 mg/kg).

Block Technique:

At the end of the surgical procedure, while patients are still under general anesthesia, the patient's envelope which contains the number of group will be opened and it will be recorded in the data collection sheet as a number of group because the data collector will be blind to the intervention which will be done to the patient, only the anesthetist knows each number will be referring to which intervention.

I) Group I (ESP Group): will receive US-guided ESPB. II) Group II (AQL Group): will receive US-guided SAQLB. III) Group III (Control Group): will receive IV multimodal analgesia only. Block techniques will be performed under complete aseptic precautions.

Time of Performing the Block:

It will be recorded and defined as the time from placement of US probe on the patient's skin till the end of local anesthetic (LA) injection. It represents the time needed for adequate ultrasonic visualization, needle introduction and drug injection. The time for skin preparation, draping, and probe sheathing will not be included.

Recovery from General Anesthesia:

After completion of blockade, isoflurane will be discontinued, residual neuromuscular blockade will be antagonized using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg) administered IV, and the patient will be extubated.

Block Assessment:

After recovery from general anesthesia, sensory blockade will be confirmed on both sides at the level of T6 dermatomal level (at the level of the xiphoid process) 30 min. after LA injection at PACU by pin prick using Hollmen scale for sensory block, as follows; 1 = Normal sensation of pinprick, 2 = Pin prick felt as sharp pointed but weaker when compared with unblocked area, 3 = Pin prick felt as touch with blunt object, 4 = No perception of pin prick. Cases of failed block, who would have Hollmen sensory scale of 1 , will be excluded from the study.

C. Postoperative Management:

Multimodal Analgesia:

Postoperative pain in the post-anesthesia care unit (PACU) and on the ward will be treated with a combination of IV multimodal analgesia in the form of Acetaminophen (15 mg/kg 4/day) and Ketorolac (0.5 mg/kg 3/day) using a fixed scheme. In addition, Nalpuphine, as 3 mg IV bolus at each dose, will be given when Numerical Rating Scale (NRS) ≥ 3. VAS will be assessed 5 - 10 min. after each opioid dose to assess the need for additional opioid doses.

Measured Parameters:

1. Time of Performing the Block.
2. Postoperative Hemodynamics; including; heart rate (HR), mean arterial blood pressure (MAP), respiratory rate (RR), and oxygen saturation (SpO2) will be recorded immediately postoperative, then every hour for the first 4 hrs, and then every 4 hrs till the end of the first 24 hrs postoperative.
3. Postoperative Pain;

   A. Patients will be instructed how to represent their level of pain using NRS 0 to 10, 0 indicated no pain, and 10 indicated the most intense pain. Taking the procedures of laparoscopic cholecystectomy (LC) into account, pain assessment was performed in four domains: pain when coughing, pain at rest, incision pain and visceral pain. Specific questions were used respectively:

   "What is NRS pain scores when you cough?" "What is your NRS pain scores when you lay down in a quiet situation?" "What is your NRS pain scores on the incision site?" "What is your NRS pain scores about dull pain inside the abdomen?" NRS will be recorded by the data collector who will be blind to the intervention done to the patient. Pain assessment will be done 30 min. postoperative, then at 2, 4, 6, 8, 12, 18 and 24 hrs postoperative.

   B. Shoulder pain (SP) will be assessed using a 3 point scale (0 = none, 1 = mild and 2 = severe) at the same time points.
4. Time of Postoperative First Opioid Analgesic Request.
5. Total Opioid Consumption in the First 24 hrs Postoperative.
6. Time To Recovery Of Intestinal Function; defined as time from recovery to first flatus.
7. Time To First Ambulation; defined as time from T0 until the subject was able to stand up and walk without support.
8. Patient Satisfaction; will be also considered and recorded at the end of the first 24 hrs postoperative using a 5-point scale of "completely dissatisfied" to "completely satisfied" as follows; 1 = Completely dissatisfied, 2 = Dissatisfied, 3 = Neither satisfied, nor dissatisfied, 4 = Satisfied, 5 = Completely satisfied.

Complications:

1. Pain:
2. Undesirable Effects of Opioid Usage; A. Sedation: will be measured using Pasero opioid-induced sedation scale (POSS); S; Sleep, easy to arouse, 1; Awake and alert, 2; Slightly drowsy, easily aroused, 3; Frequently drowsy, arousable, drifts off to sleep during conversation, 4; Somnolent, minimal or no response to verbal and physical stimulation.

   B. Respiratory Depression: defined as decreased respiratory rate (RR) < 8-10 breaths/minute or decreased oxygen saturation (SpO2) < 90%.

   Naloxone will be administered in case of excessive sedation and/or respiratory depression. Times of excessive sedation or respiratory depression, and total requirements of naloxone reversal in the first 24 hrs postoperative will be recorded.

   C. Postoperative Nausea and Vomiting (PONV): will be measured using a categorical scoring system; 0 = none, 1 = mild, 2 = moderate, 3 = severe. Detection of nausea will be occurred when nausea score > 0 at any time point postoperatively. Ondansetron (4 mg) will be administered IV in case of nausea and/or vomiting. Frequency of PONV and total requirements of ondansetron in the first 24 hrs postoperative will be recorded.
3. Technical Complications; Include visceral injury, hematoma formation, lower extremity weakness and local anesthetic systemic toxicity (LAST).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 60 years, of both sexes.
2. ASA class II - III.
3. Scheduled to undergo laparoscopic cholecystectomy under general anesthesia.
4. Body mass index (BMI) ≥ 30 kg/m².

Exclusion Criteria:

1. Age < 18 or > 60 years. 2. ASA IV patients. 4. Intraoperative conversion to open surgery. 5. Contraindications of regional anesthesia, e.g., allergy to local anesthetics, coagulopathy or infection at the site of injection.

6. Uncooperative patients or psychiatric disorders. 7. Spinal deformity or previous spine surgery. 8. Chronic use of analgesics or drug dependence. chronic pain characterized by opioid use for > 30 consecutive days within the 3 preoperative months at a dose equivalent to at least 15 mg of morphine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
24 hours Postoperative Total Opioid Consumption. | First 24 hours Postoperative
  24 hours Postoperative Total Opioid Consumption.

SECONDARY OUTCOMES:
Time of Performing the Block. | Intraoperative (Time from placement of US probe on the patient's skin till the end of local anesthetic injection.)
  Time from placement of US probe on the patient's skin till the end of local anesthetic injection.
Time of Postoperative First Opioid Analgesic Request. | First 24 hours Postoperative
  Time of Postoperative First Opioid Analgesic Request.
Postoperative NRS Scores | First 24 hours Postoperative
  NRS scores recorded 30 min. postoperative, then at 2, 4, 6, 8, 12, 18, and 24 hrs postoperative, during rest and movement.
Postoperative Complications | First 24 hours Postoperative
  including sedation, respiratory depression, PONV, visceral injury, hematoma formation, lower extremity weakness, and LAST.
Time to First Ambulation. | First 24 hours Postoperative
  time until the subject was able to stand up and walk without support.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf A Torki, MD, Principal Investigator — Anesthesia and surgical intensive care, zagazig university, faculty of medicine; Mona A Shahin, MD, Study Director — Anesthesia and surgical intensive care, zagazig university, faculty of medicine
Locations (1):
- Zagazig university hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melnyk M, Casey RG, Black P, Koupparis AJ. Enhanced recovery after surgery (ERAS) protocols: Time to change practice? Can Urol Assoc J. 2011 Oct;5(5):342-8. doi: 10.5489/cuaj.11002. PMID 22031616
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, MacFie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):783-800. doi: 10.1016/j.clnu.2012.08.013. Epub 2012 Sep 28. PMID 23099039
- [Background] Børglum J, Jensen K, Moriggl B, Lönnqvist P, Christensen AF, Sauter A and Bendtsen TF: Ultrasound-guided transmuscular quadratus lumborum blockade. Br J Anesth 2013;110 (3):297-300.
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Ahmad S, Kendall MC, McCarthy RJ. Dexamethasone to prevent postoperative nausea and vomiting: an updated meta-analysis of randomized controlled trials. Anesth Analg. 2013 Jan;116(1):58-74. doi: 10.1213/ANE.0b013e31826f0a0a. Epub 2012 Dec 7. PMID 23223115
- [Background] Peng PW, Sandler AN. A review of the use of fentanyl analgesia in the management of acute pain in adults. Anesthesiology. 1999 Feb;90(2):576-99. doi: 10.1097/00000542-199902000-00034. No abstract available. PMID 9952166
- [Background] Carassiti M, Cappiello D, Galli B. One shot six centres: a new strategy in ultrasound guided paravertebral block. J Anesth Clin Res. 2015;6: 580 - 583. doi:10.4172/2155-6148.1000580
- [Background] Capogna G, Celleno D, Laudano D, Giunta F. Alkalinization of local anesthetics. Which block, which local anesthetic? Reg Anesth. 1995 Sep-Oct;20(5):369-77. PMID 8519712
- [Background] Caljouw MA, van Beuzekom M, Boer F. Patient's satisfaction with perioperative care: development, validation, and application of a questionnaire. Br J Anaesth. 2008 May;100(5):637-44. doi: 10.1093/bja/aen034. Epub 2008 Mar 12. PMID 18337271
- [Background] Pasero C. Assessment of sedation during opioid administration for pain management. J Perianesth Nurs. 2009 Jun;24(3):186-90. doi: 10.1016/j.jopan.2009.03.005. No abstract available. PMID 19500754
- [Background] Fitzgibbon DR and McQuay H. Respiratory Depression: Incidence, Diagnosis, and Treatment. In: Sinatra RS, de Leon-Cassasola OA, Viscusi ER, Ginsberg B, editors. Acute Pain Management. Cambridge: Cambridge University Press; 2009. p. 416-30.
- [Background] Chen CK and Phui VE. The efficacy of ultrasound-guided oblique subcostal transversus abdominis plane block in patients undergoing open cholecystectomy. Southern African Journal of Anaesthesia and Analgesia. 2011;17(4):308-10.